CLINICAL TRIAL: NCT02116816
Title: Investigation Into Polyphenol Absorption Profiles
Brief Title: Absorption Profiles of Three Polyphenol Preparations With and Without Pollen Shell Covering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Protocol Version 2
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Polyphenols Absorption Profile
MeSH Terms: interventions — Polyphenols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Polyphenol (Experimental): Polyphenol preparations
  Interventions: Dietary Supplement: Polyphenol

INTERVENTIONS:
Dietary Supplement: Polyphenol — Polyphenol

SUMMARY:
This study consists of two parts. The first part of the study looked at the absorption of three different polyphenol preparations into the blood, the variability of their absorption and whether their absorption could be enhanced by mixing with pollen shells. For this purpose 12 healthy volunteers were recruited. All participants received all the 3 supplements with and without mixing with pollen shells so they had a total of 3 tests. For each test six blood samples were taken over an 8 hour period. Urine samples were also collected.

Oligopin was selected from the first study. The second part of study aims to look at the effects of Oligopin on endothelial function by assessing vascular tone and function in healthy volunteers using a non-invasive, direct measurement of vasodilatory capacity (EndoPAT). Nitrate and nitrite measurements, as well as blood pressure measurements, will also be recorded to provide a clear clinical assessment of the effects of this preparation (if any) upon vascular function. The effects of Oligopin will be compared to a placebo (methylcellulose-filled capsules) to allow a robust assessment of any clinical effects. A total of 24 healthy volunteers will be recruited for this study.

DETAILED DESCRIPTION:
This study consists of two parts. The first part of the study looked at the absorption of three different polyphenol preparations into the blood, the variability of their absorption and whether their absorption could be enhanced by mixing with pollen shells (pollen shells have been shown to enhance lipid molecule absorption). For this purpose 12 healthy volunteers were recruited. All participants received all the 3 supplements with and without mixing with pollen shells so they had a total of 3 tests. For each test six blood samples were taken over an 8 hour period. Urine samples were also collected.

Oligopin was selected from the first study. The second part of study aims to look at the effects of Oligopin on endothelial function by assessing vascular tone and function in healthy volunteers using a non-invasive, direct measurement of vasodilatory capacity (EndoPAT). Nitrate and nitrite measurements, as well as blood pressure measurements, will also be recorded to provide a clear clinical assessment of the effects of this preparation (if any) upon vascular function. The effects of Oligopin will be compared to a placebo (methylcellulose-filled capsules) to allow a robust assessment of any clinical effects. A total of 24 healthy volunteers will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects between the age of 18-65 who can speak and understand English
2. No concomitant medication including herbal medicines and food supplements
3. No concomitant disease processes
4. Body Mass Index 21- 29kg/m2
5. Systolic blood pressure ≤150 mm Hg and diastolic pressure <90 mm Hg
6. Subjects who have given informed consent

Exclusion Criteria:

1. Patients not wishing to allow disclosure to their GPs.
2. Concomitant medication including herbal medicines and food supplements
3. Concomitant disease processes
4. History of drug/alcohol abuse or Alcohol intake within 24 hours of dosing visit (visits 2-4)
5. Body Mass Index <21 and > 29kg/m2
6. Systolic blood pressure >150 mm Hg and or a diastolic pressure>90 mm Hg
7. Unable to tolerate polyphenol products or adhere to low polyphenol diet
8. Vegetarian
9. Subjects not willing or able to fast until 12 noon (a total of 14 hours).
10. Pregnant females or planning to conceive in the next 3 months.
11. Participation in any other study currently or in the last three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Absorption Curve for each polyphenol preparation | 8 hours
  Blood samples will be withdrawn 6 times over an 8 hour period: baseline, then 30 minutes, 1 hour, 2 hours, 4 hours and 8 hours after ingestion of each polyphenol supplement (total 3 supplements)

CONTACTS AND LOCATIONS:
Overall Officials: Thozhukat Sathyapalan, MBBS FRCP MD, Principal Investigator — University of Hull
Locations (1):
- Michael White Centre for Diabetes and Endocrinology, Hull, East Yorkshire, United Kingdom